CLINICAL TRIAL: NCT05699772
Title: Expanding Delivery of an Evidence-based Weight-loss Intervention to Enhance Access and Reach Underserved Groups After TBI
Acronym: tGLB-TBI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: North Texas Traumatic Brain Injury Model System (NTX-TBIMS) (Unknown); National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Evan Elizabeth Rainey, Manager, Baylor Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BSW IRB #022-356
Record Dates: First submitted 2023-01-13; First posted 2023-01-26 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Whole-Body Irradiation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth GLB-TBI (tGLB-TBI) (Experimental): The goal of the tGLB-TBI program is to help the participant achieve and maintain a 5-7% weight-loss using a two-pronged approach:
  1. Physical activity: This is based upon recommendations by the American Heart Association and the American College of Sports Medicine (ACSM) to achieve 150 minutes of moderate intensity activity each week. Walking is the primary activity recommended.
  2. Healthy eating: Based on United States Department of Agriculture guidelines, the GLB emphasizes healthy eating patterns and tracking dietary intake.
  The tGLB-TBI was modified from the DPP-GLB and is a one-year program with 22 sessions. It begins with 12 weekly sessions called the Core Program, followed by a Transition phase consisting of 2 bi-weekly and 2 monthly sessions, and a Support Phase consisting of 6 monthly sessions. Sessions will be delivered in a group setting via telehealth (Microsoft Teams).
  Interventions: Behavioral: Telehealth-delivered Group Lifestyle Balance for people with TBI (tGLB-TBI)
- Brain Health Group (BHG) (Active Comparator): The Brain Health Group (BHG) meets at the same frequency as the GLB-TBI (i.e., 22 group-based sessions, 12 weekly, 4 bi-monthly, and 6 monthly).The focus of the BHG is on brain health education, self-management, and problem-solving and the BHG did not receive any education on weight-loss strategies. Sessions will be delivered in a group setting via telehealth (Microsoft Teams).
  Interventions: Behavioral: Brain Health Group (BHG)

INTERVENTIONS:
Behavioral: Telehealth-delivered Group Lifestyle Balance for people with TBI (tGLB-TBI) — The GLB-TBI was modified from the Diabetes Prevention Program Group Lifestyle Balance (DPP-GLB) by a group of stakeholders using a community based participatory research approach. The GLB-TBI is modified for people with Traumatic Brain Injury and addresses their unique weight loss and healthy lifestyle needs.
  Arms: Telehealth GLB-TBI (tGLB-TBI)
Behavioral: Brain Health Group (BHG) — The BHG was developed by researchers and clinicians at Baylor Scott & White Institute for Rehabilitation.
  Arms: Brain Health Group (BHG)

SUMMARY:
The goal of this clinical trial is to extend the accessibility of the Diabetes Prevention Program Group Lifestyle Balance (DPP-GLB) modified for people with TBI (GLB-TBI) to reduce health inequities and reach a broad and diverse sample.

To increase the accessibility and reach of the GLB-TBI we will conduct a randomized control trial (RCT) to assess intervention efficacy of telehealth delivery of the GLB-TBI (tGLB-TBI). Results will provide a scalable telehealth weight-loss program that clinicians and community workers across the country can use to help people with TBI lose weight and improve health.

DETAILED DESCRIPTION:
Diabetes Prevention Program Group Lifestyle Balance Program (DPP-GLB): The DPP-GLB is a 12-month, evidence-based, CDC-accredited weight-loss intervention designed for delivery in group-based, community settings, and has resulted in weight loss in a variety of settings such as community centers, churches, worksites, and healthcare settings. Alternate modes of delivery (e.g., DVD, telehealth, telephone call) have also proven efficacious. The primary goal of the DPP-GLB intervention is to help the participant achieve and maintain a 5-7% weight loss by following federal guidelines for physical activity participation (safe and progressive increase to achieve 150 minutes of moderate intensity activity each week) and dietary recommendations.

DPP-GLB for individuals with TBI: In 2015 we modified the DPP-GLB with a group of stakeholders to meet the unique needs of individuals with TBI (GLB-TBI). We pilot tested the GLB-TBI in a group of 18 individuals with TBI who lost -10.2±13lbs (-5% weight-loss) over 12 months. These results warranted rigorous testing.

Efficacy of the GLB-TBI using an RCT: We then completed an in-person randomized controlled trial (RCT) to assess the efficacy of the GLB-TBI compared to an attention control (NCT03594734) for Dallas residents after TBI. Individuals in the GLB-TBI group (n=27) lost -17.8±41.4lbs (-7.9%) over the 12-month program and the attention control group (n=28) lost 0±55.4lbs (0%). The GLB-TBI group also had significant improvements in diastolic blood pressure, waist circumference, triglycerides, and HDL cholesterol. As a result of this strong evidence, our GLB-TBI curriculum was recognized by the CDC as an evidence-based approach to in-person weight-loss.

The goal of this clinical trial is to extend the accessibility of the Diabetes Prevention Program Group Lifestyle Balance (DPP-GLB) modified for people with TBI (GLB-TBI) to reduce health inequities and reach a broad and diverse sample.

To increase the accessibility and reach of the GLB-TBI we will conduct a randomized control trial (RCT) to assess intervention efficacy of telehealth delivery of the GLB-TBI (tGLB-TBI). Results will provide a scalable telehealth weight-loss program that clinicians and community workers across the country can use to help people with TBI lose weight and improve health.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age
* Greater than or equal to 6 months post traumatic brain injury (TBI)
* Moderate to severe TBI at time of injury
* Body Mass Index greater than or equal to 25
* Able to participate in physical activity
* Willing to use a tablet/computer/smartphone (either personal device or one provided by the research team)

Exclusion Criteria:

* Contraindications to physical activity (e.g., uncontrolled hypertension, unstable angina, severe joint disease, uncontrolled vertigo/dizziness)
* Not fluent in the English language
* Low cognitive function
* Residing in a hospital, acute rehabilitation facility, or skilled nursing facility
* Diagnosed with or taking medications for Type 2 diabetes
* Self-reported pregnancy
* Pre-existing diagnosis of an eating disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Weight | Baseline, 3, 6, and 12 months
  Weight will be obtained at a lab local to the participant based on their preference. Weight for participants randomized to the GLB-TBI will also be captured via self-weighing using provided BodyTrace Smart Scale, which include cellular connectivity so weight will be sent directly to the research team. The scales have demonstrated good concordance rates with in-person weighing in previous weight management research.Scales will be setup by our team before being mailed to participants with instructions for use.

SECONDARY OUTCOMES:
Change in Hemoglobin A1c (HbA1c) | Baseline, 3, 6, and 12 months
  Hemoglobin A1c will be obtained at a lab local to the participant based on their preference.
Change in Lipid Panel | Baseline, 3, 6, and 12 months
  Total cholesterol, HDL, LDL, and triglycerides will be obtained at a lab local to the participant based on their preference
Change in Arm Circumference | Baseline, 3, 6, and 12 months
  Arm circumference will be measured at the mid-upper arm at a lab local to the participant based on their preference.
Change in Waist Circumference | Baseline, 3, 6, and 12 months
  Waist circumference will be measured at the umbilicus at a lab local to the participant based on their preference.
Change in Blood Pressure | Baseline, 3, 6, and 12 months
  Measured using an automatic cuff (average of three readings, patient seated) diastolic and systolic scores will be recorded at a lab local to the participant based on their preference.
Change in 8-Year Diabetes Risk | Baseline, 3, 6, and 12 months
  The Framingham Heart Study diabetes risk score will be calculated using predictors including age, gender, fasting glucose, BMI, HDL cholesterol and triglyceride levels, blood pressure, and parental history. Risk score calculator and regression model are free and used in GLB weight-loss trials.
Change in Metabolic Syndrome Severity Score | Baseline, 3, 6, and 12 months
  Metabolic Syndrome is a cluster of cardiovascular risk factors that include abdominal obesity (large waist circumference, high BMI), high blood pressure, high triglycerides, low HDL cholesterol and high fasting blood sugar. Individuals who have ≥3 of these risk factors have metabolic syndrome, placing them at greater risk of developing heart disease and diabetes. As metabolic syndrome is sensitive to lifestyle change, the metabolic syndrome severity score calculator is used to determine risk for future cardiovascular disease compared to the US population. Risk scores below 0 indicate a lower degree of metabolic syndrome risk than the average US adult; scores above 0 are associated with greater risk for disease. A score of 1 indicates risk is higher than 84.1% of US adults and a score of 2 is higher than 97.7% of US adults. Z scores are calculated for BMI and waist circumference.
Change in Dietary Change | Baseline, 3, 6, and 12 months
  The DPP-GLB program itself utilizes food logs as an intervention behavioral tool, however, to further evaluate intervention efficacy we will also assess dietary change at each assessment period. 24-hour dietary recalls will be collected with the latest version of the Automated Self-Administered 24-hour (ASA24) Dietary Assessment Tool 1-day prior to the telephonic follow-up. This free online platform (https://epi.grants.cancer.gov/asa24/#what; uses interactive multi-pass methodology68(gold-standard in dietary assessment) and provides an overall diet quality score, the Healthy Eating Index (available online through the NCI website [https://epi.grants.cancer.gov/asa24/resources/hei.html] and aligns with federal recommendations and guidelines).
Change in Neighborhood Environment Walkability Scale (NEWS) | Baseline, 3, 6, and 12 months
  The Neighborhood Environment Walkability Scale (NEWS) assesses participants' perception of neighborhood features related to physical activity and grocery shopping, including residential density, land use mix (including both indices of proximity and accessibility), street connectivity, infrastructure for walking/cycling, neighborhood aesthetics, traffic and crime safety, and neighborhood satisfaction. Questions are rated on a 4-point Likert scale with higher scores signifying greater perceived walkability. Scores provide insight into environmental barriers faced, are sensitive to behavior change, and can be used as a covariate for weight-loss. This measure will be delivered telephonically.
Change in Healthy Eating and Physical Activity | Baseline, 3, 6, and 12 months
  The Behavioral Risk Factor Surveillance System (BRFSS) is a state-based system of health surveys that collects information on health risk behaviors, preventative health practices, and health care access primarily related to chronic disease and injury. The GLB-TBI uses the two subscales of Healthy Eating and Physical Activity from the 2017 version of the BRFSS. It consists of 14 items. For this study, we will capture minutes of self-reported physical activity (higher numbers signify more physical activity and better outcome) and number of whole fruits/vegetables consumed each day (higher numbers mean better outcome). This measure will be administered telephonically.
Change in Self-Rated Abilities for Health Practice (SRAHP) | Baseline, 3, 6, and 12 months
  The SRAHP includes 28 items to assess health behaviors among people with disabilities and yields a total Health Practices Score plus 4 subscale scores (Exercise, Nutrition, Health Practices, and Psychological Well Being). Items are rated on a 5-point scale from 0 'not at all' to 4 'completely.' Scores range from 0-28 with higher scores indicating higher self-efficacy for the health behaviors. This measure will be administered telephonically.
Change in Quality of Life After Brain Injury - Overall Scale | Baseline, 3, 6, and 12 months
  The Quality of Life After Brain Injury - Overall Scale (QOLIBRI-OS) is a six-item self-report questionnaire addressing how satisfied individuals are with aspects of their functioning (physical; cognitive; emotional; participation; social life; future prospects). Answers are on a 5-point Likert scale and the sum of all items are converted to a percentage scale from 0-100. The QOLIBRI-OS has excellent reliability and internal consistency. This measure will be administered telephonically.
Change in Telehealth Usability Questionnaire (TUQ) | Baseline, 3, 6, and 12 months
  The Telehealth Usability Questionnaire (TUQ) is a validated assessment that measures 5 usability factors of telehealth (usefulness, ease of use, effectiveness, reliability, and satisfaction). 21 items are scored on level of agreement from 1-7, with higher scores indicating greater agreement. All subscales have good to excellent reliability (α=.79-.92). This measure will be administered telephonically.
Change in Exit Survey | 12 months
  Participants will be asked to complete an exit survey at the 12-month assessment. This survey will ask about participant experience in, and satisfaction with, the GLB-TBI telehealth program and suggestions for improvement. The survey will be emailed to participants via a secure link.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Driver, PhD, Principal Investigator — Baylor Research Institute
Locations (1):
- Baylor Scott & White Research Institute, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
IPD requests can be made to the Principal Investigator via email (Evan.McShan@BSWHealth.org).